CLINICAL TRIAL: NCT03259685
Title: Effect of Free Sugar Replacement With Non-nutritive Sweeteners on Metabolic Health of High Sugar Sweetened Beverages Consumers: Potential Role of the Gut Microbiome
Brief Title: Effect of Non-nutritive Sweeteners of High Sugar Sweetened Beverages on Metabolic Health and Gut Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Marie-Claude Vohl, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SBG 2017-136
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gut Microbiota; Metabolic Syndrome
Keywords: Non-nutritive sweeteners; High Sugar Sweetened Beverages; Diet
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular beverages (Active Comparator): Sugar sweetened soft drinks
  Interventions: Other: 710 ml of regular soft drinks, taken daily for 10 weeks
- Diet beverages (Experimental): Soft drinks sweetened with artificial non-nutritive sweeteners (i.e. aspartame, acesulfame-K)
  Interventions: Other: 710 ml of diet soft drinks, taken daily for 10 weeks
- Stevia beverages (Experimental): Soft drinks sweetened with natural non-nutritive sweeteners (i.e. steviol glycosides)
  Interventions: Other: 710 ml of stevia-sweetened soft drinks, taken daily for 10 weeks

INTERVENTIONS:
Other: 710 ml of regular soft drinks, taken daily for 10 weeks — Subjects will consume regular soft drinks to test if there is a significant difference on the impact on gut microbiota composition and metabolic syndrome parameters between this treatment and the active treatments (diet and stevia beverages).
  Arms: Regular beverages
Other: 710 ml of diet soft drinks, taken daily for 10 weeks — Subjects will consume diet soft drinks during 10 weeks to test the possible effects of aspartame/acesulfame-K sweetened beverages on gut microbiota composition and on metabolic syndrome parameters.
  Arms: Diet beverages
Other: 710 ml of stevia-sweetened soft drinks, taken daily for 10 weeks — Subjects will consume soft drinks containing stevia during 10 weeks to test the possible effects of steviol glycosides sweetened beverages on gut microbiota composition and on metabolic syndrome parameters.
  Arms: Stevia beverages

SUMMARY:
Increasing evidence suggest that artificial sweeteners such as saccharin, aspartame and sucralose may not be as metabolically safe as they first appeared, and it has been proposed that their consumption may be linked to important disturbances in the gut microbiome. Some in vitro and in vivo studies suggest that the recently approved sugar substitute Stevia (eg. steviol glycosides) can also influence intestinal homeostasis. However, it is not clear whether this natural non-nutritive sweetener (NNS) could also cause metabolic and microbiome disturbances as proposed for their synthetic counterparts. In fact, steviol glycosides may even have a beneficial impact on glucose homeostasis and lipid metabolism possibly through a positive action on intestinal health and gut microbiome, but this has yet to be experimentally tested in a rigorous study.

The main objective of this project is to evaluate whether steviol glycosides sweetened beverages (SGSB) or aspartame/acesulfame K sweetened beverages (AASB) exert beneficial, neutral or detrimental effects on metabolic health of regular consumers of sugar-sweetened beverages (SSBs), and whether modulation of the gut microbiome is involved in the resulting impact of these NNSs on metabolic health.

As chronic overconsumption of SSBs is clearly associated with an increased cardiometabolic risk, this study will be the first to determine the metabolic impact of replacing SSBs by potentially "healthier alternatives" such as the increasingly popular stevia-based soft drinks and aspartame-based soft drinks. The investigators will further investigate whether these NNS can cause pernicious effects on intestinal health and the gut microbiome. It is a crucial concern since the importance of this unsuspected key "organ" has been ignored for too long and its important implication in many chronic societal diseases has just been discovered.

Results of this study could have a direct influence on health, nutrition and even agricultural policies as well as dietary guidelines around the world. This project is also critically important as an increasing amount of health professionals such as physicians, nurses and registered dietitians seek to provide evidenced-based guidance to individuals looking for healthier alternatives to SSBs including stevia-based or aspartame-based soft drinks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women in good health
* Soft drinks consumers (between 4 cans/week to 4 cans/day)

Exclusion Criteria:

* Metabolic disorders (hypertension, diabetes, hypercholesterolemia)
* Daily consumption of more than 4 cans of soft drinks
* Regular use of medication affecting study parameters
* Change of medication (type or dose) in the last year
* Use of antibiotics in the last 3 months
* Change in natural health product use in the last 3 months
* More than 2 alcohol drinks par day
* Weight change of more than 5% in the last 3 months
* Surgery in the last 3 months or planed during the study
* Allergy or intolerance for products contained in soft drinks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolic syndrome parameters including insulin/glucose homeostasis and lipid/lipoprotein metabolism in sugar-sweetened beverages (SSB) consumers following regular, diet or stevia-sweetened beverages intakes for 10 weeks. | 18-24 months

SECONDARY OUTCOMES:
Changes in intestinal homeostasis of SSB consumers following regular, diet or stevia-sweetened beverages intakes for 10 weeks. | 4-6 months
Changes in gut microbiota composition of SSB consumers following regular, diet or stevia-sweetened beverages intakes for 10 weeks. | 4-6 months

OTHER OUTCOMES:
Changes in key molecular signaling pathways and metabolic regulatory networks identified through transcriptomics and metabolomics of SSB consumers following regular, diet or stevia-sweetened beverages intakes for 10 weeks. | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Vohl, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada

REFERENCES:
- [Derived] Bergwall S, Johansson A, Sonestedt E, Acosta S. High versus low-added sugar consumption for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2022 Jan 5;1(1):CD013320. doi: 10.1002/14651858.CD013320.pub2. PMID 34986271